CLINICAL TRIAL: NCT00012584
Title: A Treatment Study of Youth With Comorbid Attention Deficit Hyperactivity Disorder (ADHD) and Anxiety Disorders
Brief Title: Treatment of Youth With ADHD and Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: N01MH12012 (NIH); DSIR CT
Record Dates: First submitted 2001-03-14; First posted 2001-03-16 (Estimated); Last update posted 2009-06-24 (Estimated); Status verified 2009-06

CONDITIONS: Attention Deficit Hyperactivity Disorder; Anxiety, Separation; Social Phobia; Generalized Anxiety Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Anxiety, Separation; Phobia, Social; Generalized Anxiety Disorder | interventions — Methylphenidate; Fluvoxamine

INTERVENTIONS:
Drug: methylphenidate
Drug: fluvoxamine

SUMMARY:
The purpose of this NIMH-sponsored pilot study is to collect information on the efficacy and safety of drug treatments for children and adolescents who suffer from both ADHD and anxiety disorders. Specifically, the study will examine the benefits of the stimulant medication both alone and in combination with fluvoxamine, a selective serotonin reuptake inhibitor (SSRI) that has antianxiety effects. Young people aged 6 to 17 diagnosed with these co-occurring disorders may be eligible to participate.

DETAILED DESCRIPTION:
Many children and adolescents with mental disorders in the United States are treated with multiple psychotropic medications even though there is not much information on how well these medications work together or if they are safe to administer together. Many youth with ADHD have co-occurring (comorbid) disorders such as oppositional-defiant disorder, anxiety disorders, and mood disorders. There is much interest in the treatment of children and adolescents with comorbid ADHD and anxiety disorders because this is a common condition in clinical practice. When children with both anxiety and ADHD receive stimulant medication for ADHD, their anxiety may not improve. SSRI medications represent a reasonable addition to stimulant treatment, as they are considered effective for anxiety disorders based on controlled trials in adults and open trials in children. However, there are no data from controlled studies regarding the tolerability and dosing of the combination of stimulant treatment (including methylphenidate) and SSRIs in the treatment of children with comorbid ADHD and anxiety disorder.

In this study, children and adolescents will be evaluated for the presence of both ADHD and Anxiety Disorder. Approximately 120 children and adolescents with both disorders who meet all the study entry requirements (such as being otherwise medically healthy) will be enrolled. Children and adolescents who are not on a stable dose of a stimulant will first be treated openly with methylphenidate for 6 weeks. Those whose ADHD does not improve during this initial treatment period will not continue in the study but will be referred for further support in the community. Those who show improvement in both their ADHD and anxiety symptoms will stay on methylphenidate for an additional 8 weeks. Those who show improvement in ADHD but not anxiety will be asked to enter the double-blind phase of the study. In this phase, participants will be randomized (assigned by chance) to receive either fluvoxamine or placebo, in combination with stimulant/methylphenidate, for 8 weeks. Children or adolescents who enter the study on a stable dose of stimulant will move directly to the Double-Blind phase. Participants who are assigned to placebo and who do not show an improvement in anxiety after 8 weeks will be eligible for an additional 8 weeks of open treatment with the methylphenidate/stimulant and fluvoxamine combination. At the end of the trial, clinical care will be provided for up to an additional month until referral to an outside clinician can be arranged.

ELIGIBILITY:
* ADHD diagnosis
* DSM-IV diagnosis of anxiety
* IQ greater than 70
* residence with primary caretaker for at least 6 months
* ages 6-17 and attending school
* no previous treatment failure to or intolerance of fluvoxamine or methylphenidate (unless currently taking another stimulant)

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120
Dates: Start 2000-11; Primary Completion 2002-05 (Actual); Study Completion 2002-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - UCLA Neuropsychiatric Institute, Los Angeles, California
  - Johns Hopkins School of Medicine, Baltimore, Maryland
  - New York University Child Study Center, New York, New York
  - New York State Psychiatric Institute, New York, New York
  - Duke University Medical Center, Durham, North Carolina

REFERENCES:
- [Background] Fluvoxamine for the treatment of anxiety disorders in children and adolescents. The Research Unit on Pediatric Psychopharmacology Anxiety Study Group. N Engl J Med. 2001 Apr 26;344(17):1279-85. doi: 10.1056/NEJM200104263441703. PMID 11323729
- [Background] Coyle JT. Drug treatment of anxiety disorders in children. N Engl J Med. 2001 Apr 26;344(17):1326-7. doi: 10.1056/NEJM200104263441711. No abstract available. PMID 11320394
- See also: More information on ADHD — http://www.nimh.nih.gov/health/topics/attention-deficit-hyperactivity-disorder-adhd/index.shtml
- See also: More information on anxiety — http://www.nimh.nih.gov/health/topics/anxiety-disorders/index.shtml